CLINICAL TRIAL: NCT02583087
Title: Endoscopic Submucosal Dissection for the Treatment of Early Barrett's Neoplasia
Brief Title: ESD for the Treatment of Early Barrett's Neoplasia
Acronym: ESTEBAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hôpital Cochin (Other)
Collaborators: French Society of Digestive Endoscopy (Other); European Georges Pompidou Hospital (Other); Hôpital Edouard Herriot (Other); Hospital Prive Jean Mermoz (Other); University Hospital, Limoges (Other); University Hospital, Bordeaux (Other); Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Principal Investigator, Frederic PRAT, Professor Frederic Prat, Hôpital Cochin
Other Study IDs: 20102015
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Barrett Esophagus; Esophageal Neoplasm
Keywords: Barrett esophagus; Esophageal adenocarcinoma; Endoscopic submucosal dissection
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms; Adenocarcinoma Of Esophagus | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: endoscopic submucosal dissection — Endoscopic resection of a superficial neoplastic lesion of the esophagus, including the mucosal and the submucosa resected en bloc.
  Other Names: endoscopic resection; ESD

SUMMARY:
This study assesses the quality of the resection of early neoplasia arinsing in Barrett's esophagus using endoscopic submucosal dissection. It is a multicenter prospective registry among 7 centers including all consecutive patients with early Barrett's neoplasia of 15 mm or more in size treated by endoscopic submucosal dissection.

DETAILED DESCRIPTION:
Endoscopic submucosal dissection ( ESD) demonstrated great efficacy in the treatment of squamous cell carcinoma of the esophagus. Results for the treatment of esophageal adenocarcinoma arising in Barrett's esophagus are conflicting.

In this multicenter prospective registry among 7 French centers, all consecutive patients with early Barrett's neoplasia of 15 mm or more in size treated by endoscopic submucosal dissection will be included in the registry. The primary objective is to assess the quality of the resection by ESD of early Barrett's neoplasia (T1A or T1B sm1 or high grade dysplasia). Secondary endpoints are to assess the combined efficacy of a treatment associating ESD and radiofrequency ablation of the remaining Barrett esophagus, and to assess the durability of the results after 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Barrett's esophagus at least C0M2 with histological documentation of intestinal metaplasia
* Visible abnormality of at least 15 mm in size
* Absence of mediastinal or coeliomesenteric enlarged lymph nodes or muscle layer invasion on pretherapeutic EUS
* Absence of mediastinal or coeliomesenteric enlarged lymph nodes or metastases on pretherapeutic CT scan

Exclusion Criteria:

* History of esophageal external irradiation
* History of esophagectomy or gastrectomy gastrectomie ou d'oesophagectomie
* Esophageal stricture
* Esophageal varices grade 3 or of any grade with signs of recent bleeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 90 years old with a visible lesion suspected of adenocarcinoma arising in a Barrett's esophagus amenable to resection by ESD.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-01-02 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Rate of histologically complete (R0) resection of esophageal adenocarcinoma or high grade dysplasia | 3 months after ESD initial procedure
  R0 resection rate = horizontal margins free from cancer or high grade dysplasia, and vertical margins free from carcinoma.

SECONDARY OUTCOMES:
Rate of en bloc resection via ESD | 3 months after ESD initial procedure
  presence of a single fragment of tissue on histopathological analysis
Rate of histologically complete (R0) resection of esophageal adenocarcinoma | 3 months after ESD initial procedure
  R0 resection rate = horizontal margins free from cancer, and vertical margins free from carcinoma.
Rate of histologically complete (R0) resection of low grade dysplasia | 3 months after ESD initial procedure
  R0 resection rate = horizontal margins free from cancer, high or low grade dysplasia, and vertical margins free from carcinoma.
Curative resection rate of adenocarcinoma | 3 months after ESD initial procedure
  R0 resection of adenocarcinoma, with submucosal invasion <500micrometers, absence of poor differenciation or lymphovascular invasion
Complication rates | 3 months
  early or late complications of ESD
rate of complete remission of adenocarcinoma, high grade dysplasia, low grade dysplasia, and intestinal metaplasia at 1 and 3 years | 3 years after initial procedure
  rate of normal endoscopic and histologic follow-up after ESD
rate of buried glands | 3 years
  Presence of Buried glands on histological analysis of follow-up biopsies

CONTACTS AND LOCATIONS:
Locations (1):
- Cochin Hospital, Paris, France